CLINICAL TRIAL: NCT06809868
Title: Role of Transposable Elements in Septic Immune Aging
Acronym: SITE
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-39420
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Sepsis and Septic Shock; Sepsis With Multiple Organ Dysfunction (MOD); Sepsis With Acute Organ Dysfunction; Sepsis, Severe; Sepsis at Intensive Care Unit; Sepsis, Severe Sepsis and Septic Shock; Sepsis, Septic Shock
Keywords: Sepsis; Transposable Elements; Immune Aging; Mortality; Secondary Infections; Critical Care Medicine (ICU)
MeSH Terms: conditions — Sepsis; Shock, Septic; Coinfection | interventions — RNA; Sequence Analysis, DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: Samples With DNA — Serum, Plasma, RNA, and DNA from patients with sepsis will be retained and analyzed as part of this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Sepsis: Adult patients (age 18 and older) admitted to the intensive care unit (ICU) meeting Sepsis 3 Criteria.
  Interventions: Genetic: RNA and DNA Sequencing
- Healthy Individual Controls: Healthy individuals not admitted to the hospital.
  Interventions: Genetic: RNA and DNA Sequencing

INTERVENTIONS:
Genetic: RNA and DNA Sequencing — DNA and RNA sequencing will be conducted on both control participants and patients with sepsis who are admitted to the ICU.

SUMMARY:
The goal of this observational study is to learn about how transposable element levels affect the patient outcomes in sepsis. The main questions it aims to answer is:

1. Do transposable elements prematurely age the immune systems of patients with sepsis?
2. Do transposable elements correlate with increased mortality in patients with sepsis in the ICU?
3. Do transposable elements correlate with increased amount of secondary infections in patients with sepsis in the ICU?

Participants will have blood drawn from them but will not be subjected to additional interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Admitted to ICU with sepsis (Sepsis 3 Criteria)
* SOFA score of at least 2 at time of enrollment

Exclusion Criteria:

* Patients on organ transplantation immunosuppression
* Patients with preexisting leukopenia
* Cancer patients receiving CAR-T therapy
* Patients who are under 18 years of age or otherwise deemed pediatric
* Patients with an ongoing bleeding diathesis (ie: DIC, hemorrhagic shock)
* Patients with a chronic hemoglobin below 7.0
* Patients who, prior to their ICU admission, are blood transfusion dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients admitted to the intensive care unit with sepsis with a SOFA score of at least 2. Sepsis is defined by the Sepsis 3 Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2028-02-14 (Estimated); Study Completion 2028-08-14 (Estimated)

PRIMARY OUTCOMES:
Immune Aging | 6 weeks

SECONDARY OUTCOMES:
Mortality (30-day) | 30 days
Secondary Infection | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexendar R Perez, M.D., Ph.D, Principal Investigator — University of California, San Francisco; Judith Hellman, M.D., Principal Investigator — University of California, San Francisco; Matthieu Legrand, M.D., Ph.D, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code